CLINICAL TRIAL: NCT05720884
Title: Efficacy and Safety of Acupuncture for Blood Pressure Fluctuation During Total Laparoscopic Hysterectomy: a Randomized Controlled, Parallel-grouped Pilot Study
Brief Title: Acupuncture for Blood Pressure Fluctuation During Total Laparoscopic Hysterectomy
Acronym: ASBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Jee Young Lee, assistant professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ICICC-CT-22-05
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Total Laparoscopic Hysterectomy
Keywords: general anesthesia; blood pressure fluctuation; acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: acupuncture group and placebo group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The intervention researcher is not blinded since the researcher should perform different intervention according to the group. However, we separate the person and location to keep the blindness as robust as possible. Both the participant and the assessor are blinded and the location where intervention is performed is separate from the location where assessment is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): A total 10 acupoints of bilateral PC6, PC5, SP3, KI3, and ST36 will be chosen for the intervention group, also known as the acupuncture group. The depth of acupuncture will be varied by participant by participant. After acupuncture needles be inserted, the needles will be manually manipulated to obtain pre-determined sensation, the De Qi. Then, acupuncture will remain inserted for 20 minutes.
  Interventions: Device: acupuncture
- placebo group (Placebo Comparator): Ten other points, which are not official acupoints and those are not on the median nerve or peroneal nerve, will be chosen for the placebo group.
  Interventions: Device: placebo acupuncture

INTERVENTIONS:
Device: acupuncture — Acupuncture of a disposable, sterilized, stainless steel needle of 0.20 mm * 30 mm size (Dongbang medical, Boryeong, Rep of Korea) will be used.
  Arms: acupuncture group
Device: placebo acupuncture — Acupuncture of a disposable, sterilized, stainless steel needle of 0.20 mm * 30 mm size (Dongbang medical, Boryeong, Rep of Korea) will be used but in differene location.
  Arms: placebo group

SUMMARY:
The goal of this pilot clinical trial is to learn about efficacy of acupuncture about blood pressure fluctuation during total laparoscopic hysterectomy in patients with uterine fibroid.

Participants will receive two times of acupuncture treatment before surgery and researchers will compare to see if acupuncture treatment would stabilize blood pressure fluctuation especially from induction time to post-incision moment.

DETAILED DESCRIPTION:
After sufficient explanation about the purpose and methods of this clinical study by a researcher, the subject who voluntarily decided to participate and signed a written consent will be evaluated for eligibility at the screening visit. Eligible subjects will be determined as acupuncture group and a placebo control group according to the randomization. Acupuncture treatment is performed twice, one day before surgery and the same day.

On the day of surgery, after entering the operating room, monitoring equipments (non-invasive blood pressure monitor, pulse oxygen saturation, electrocardiogram, anesthesia depth sensor, neuromuscular monitor) will be installed and vital signs including pulse rate, blood pressure, oxygen saturation are measured.

Anesthesia was induced with an anesthetic (intravenous propofol 1-2.5 mg/kg, IV), an analgesic (remifentanyl 0.2mg/hr, IVF), and a muscle relaxant (intravenous rocuronium 0.6-1.2 mg/kg). After induction of anesthesia, anesthesiologist performed tracheal intubation maintaining an appropriate depth of anesthesia (Sedline < 50). Mechanical ventilation started keeping end-tidal CO2 pressure of 25-35 mmHg). Then, an additional venous tube was secured. Additional disinfection process was performed, surgery is prepared.

With the patient in the lithotomy position and under the general anesthesia, the abdomen was prepared, painted and draped with the usual manner. The uterine elevator was inserted. Skin incision was performed and trocar was inserted. The CO2 gas was infused to make pneumoperitoneum which pressure was reached to 12mmHg. Entering into the abdominal cavity, the patient position was changed to the Trendelenburg position. And then the pelvic cavity and whole abdomen were examined. Bilateral pelvic side wall triangles were opened in parallel to infundibulopelvic ligament and ureter dissection was done. The ureteral course was identified, and then the right round ligament and ovarian ligament were coagulated with bipolar endocoagulator, cut with endoscissors. The left sided uterine ligaments were manipulated with the same method as above. The bladder flap was pushed and posterior broad ligament was mobilized. Bilateral uterine vessels were skeletonized and bilateral uterine vessels were coagulated and then cut. Circumferential colpotomy was done with unipolar scissor, and the uterus was removed transvaginally and then vaginal cuff was closed intracorporeal continuous suture. Hemostasis and ureteral peristalsis were assured and abdominal cavity was irrigated with normal saline. The subcutaneous tissue and the skin were closed layer by layer. In all processes, a qualified anesthesiologist whose clinical experience of more than 10 years will control the analgesic or anesthetic injection rate and inhalation gas concentration to maintain the appropriate blood pressure and depth of anesthesia.

ELIGIBILITY:
Adulthood participants who were planned to have surgical removal of uterus for uterine fibroid and have expected date of total laparoscopic hysterectomy by a gynecologist were eligible.

Inclusion criteria

1. between age of 19 and 69,
2. American Society of Anesthesiologists (ASA) class I or II,
3. required surgical removal of uterus by a gynecology specialist,
4. scheduled to have total laparoscopic hysterectomy in advance.

Exclusion criteria

1. expected survival within 3 months,
2. emergency operation which was not scheduled in advance,
3. hypertension or hypotension that can significantly interfere with the study result,
4. diagnosis of arrhythmia, such as atrial fibrillation, frequent ventricular or supraventricular premature beats,
5. diagnosis of heart failure or valvular disease,
6. anemia of hemoglobin < 12 g/dL,
7. incapable of surgery due to hemodynamic or medical reasons other than stated above,
8. incapable of receiving acupuncture treatment on determined location,
9. current use of gonadotropin-releasing hormone receptor agonists,
10. current use of drugs that may interfere with the result, including steroids, immunosuppressants, and psychiatric disorders,
11. significant comorbidities that may interfere with the interpretation of intervention efficacy or results, such as stroke, myocardial infarction, kidney disease, dementia, or epilepsy,
12. pregnant, planning to be pregnant within study period, or breastfeeding,
13. previous participation in any other clinical trial within 1 month of participation, planning to participate another clinical trial within 6 months after enrollment date, or planning to participate another clinical trial on follow-up period,
14. fail to write the informed consent form voluntarily,
15. being deemed to be unsuitable for participation.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
changes in mean blood pressure | At operation time
  the difference between the highest mean blood pressure and the lowest mean blood pressure from the induction of anesthesia to the post-incision period

SECONDARY OUTCOMES:
blood pressures according to predetermined timepoints | At operation time
  systolic blood pressure, diastolic blood pressure and mean blood pressure values at entering operation room, induction time, intubation time, venous tube insertion, preparation time, skin incision, and gas inflation.
incidence of hypotension | At the end of operation moment
  Total incidence count of hypotension events, determined as lower than 80% of baseline or systolic blood pressure below 90
incidence of hypertension | At the end of operation moment
  Total incidence count of hypertension events, determined as systolic blood pressure over 160
incidence of tachycardia according to predetermined timepoints | At the end of operation moment
  heart rate values at entering operation room, induction time, intubation time, venous tube insertion, preparation time, skin incision, and gas inflation.
incidence of bradycardia according to predetermined timepoints | At the end of operation moment
  heart rate values at entering operation room, induction time, intubation time, venous tube insertion, preparation time, skin incision, and gas inflation.
total use of remifentanil | At the end of operation moment
  Use of remifentanil dosage will be surrogate markers of stable general anesthesia.
numeric rating scale for pain | before operation(operation date), at the end of operation moment
  numeric rating scale is a 11 point scale that defined point 0 as totally painless state, and point 10 as extreme pain as imaginable as possible.
Spielberger's State-Trait Anxiety Inventory (STAI) | before operation(operation date), at the end of operation moment
  State-Trait Anxiety Inventory (STAI) consists of two categories, twenty items of questionnaire to assess state anxiety (STAI-S) and another twenty items to assess trait anxiety (STAI-T). STAI varies from a minimum score of 20 to a maximum score of 80. Lower scores means presence of less anxiety (no or low anxiety 20-37, moderate 38-44, and high anxiety 45-80).
EuroQoL-5 Dimensions - 5 Levels (EQ-5D-5L) | before operation(operation date), at the end of operation moment
  The EQ-5D-5L is used to assess effects on patients' quality of life. The questionnaire consists of questions in five areas (mobility, self-care, usual activities, pain, and anxiety/depression) that ask about the patient's current state of health. Answers are provided on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jee Young Lee, Dr, Principal Investigator — Cha Ilsan Medical Center
Locations (1):
- Lee Jee Young, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data, since researchers considered privacy.

REFERENCES:
- [Derived] Lee JY, Roh JW, Han KH, Kim MJ, Na YJ, Yun BS, Lee J. Rationale for the Use of Acupuncture to Stabilize Blood Pressure Fluctuations During Total Laparoscopic Hysterectomy: Protocol for a Pilot Parallel-Group Randomized Clinical Trial. JMIR Res Protoc. 2025 Jul 22;14:e77009. doi: 10.2196/77009. PMID 40603084